CLINICAL TRIAL: NCT00032097
Title: A Phase I Trial To Evaluate Repetitive Intravenous Doses Of Gadolinium-Texaphyrin As A Radiosensitizer In Patients With Glioblastoma Multi Forme
Brief Title: Motexafin Gadolinium in Treating Patients With Glioblastoma Multiforme Who Are Undergoing Radiation Therapy to the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069257; NABTT-2116; JHOC-NABTT-2116
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2004-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — motexafin gadolinium; Radiotherapy

INTERVENTIONS:
Drug: motexafin gadolinium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as motexafin gadolinium may make the tumor cells more sensitive to radiation therapy.

PURPOSE: Phase I trial to study the effectiveness motexafin gadolinium in treating patients with glioblastoma multiforme who are undergoing radiation therapy to the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of 2 different schedules of motexafin gadolinium as a radiosensitizer in patients with glioblastoma multiforme receiving cranial radiotherapy.
* Determine the maximum tolerated doses of this drug on these 2 schedules in these patients.
* Determine the pharmacokinetic profile of this drug in these patients.
* Determine the biodistribution of this drug in both neoplastic tissue and normal brain parenchyma in these patients.
* Determine the effect and accumulation of this drug in both normal brain parenchyma and neoplastic tissue in these patients.
* Correlate the effect and accumulation of this drug in both normal brain parenchyma and neoplastic tissue with the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter, dose-escalation study of motexafin gadolinium (PCI-0120). Patients are sequentially assigned to 1 of 2 treatment groups.

* Group I: Patients receive PCI-0120 IV over 30-60 minutes once every other day for 6 weeks. Patients concurrently undergo cranial radiotherapy once daily 5 days a week for 6 weeks.
* Group II: Patients receive PCI-0120 IV over 30-60 minutes once daily concurrently during radiotherapy. Patients undergo cranial radiotherapy as in group I.

Cohorts of 3-6 patients in each group receive escalating doses of PCI-0120 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 1 month and then every 2 months thereafter.

PROJECTED ACCRUAL: Approximately 18-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial grade IV astrocytoma

  * Glioblastoma multiforme
  * Previously untreated disease
* Measurable and contrast-enhancing tumor by MRI after incomplete resection/biopsy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT/SGPT no greater than 4 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 4 times ULN
* PT/APTT normal

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No uncontrolled hypertension

Other:

* Mini mental state exam score at least 15
* No history of glucose-6-phosphate dehydrogenase deficiency or porphyria
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of the breast
* No serious infection
* No other medical illness that would preclude study participation
* No allergy to MRI contrast (e.g., motexafin gadolinium)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy or immunotherapy for this disease, including any of the following:

  * Immunotoxins
  * Immunoconjugates
  * Antisense therapy
  * Peptide receptor antagonists
  * Interferons
  * Interleukins
  * Tumor-infiltrating lymphocytes
  * Lymphokine-activated killer cell therapy
  * Gene therapy

Chemotherapy:

* No prior chemotherapy for this disease

Endocrine therapy:

* Must be on a stable corticosteroid regimen (i.e., no increase within 5 days prior to treatment on this protocol)
* No other prior hormonal therapy for this disease

Radiotherapy:

* No prior radiotherapy for this disease

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04

CONTACTS AND LOCATIONS:
Overall Officials: James L. Pearlman, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States